CLINICAL TRIAL: NCT04826887
Title: SOLTIVE™ Laser Enucleation for Treatment of Benign Prostatic Hyperplasia
Status: Completed | Type: Observational
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Don Neff, MD, FACS, Principle Investigator, University of Kansas Medical Center
Other Study IDs: GU-EN-Solep-01
Record Dates: First submitted 2021-01-20; First posted 2021-04-01 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-09

CONDITIONS: BPH; Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Standard of Care; Lasers, Solid-State

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Solep Arm: Use of SOLTIVE Thulium Laser for HoLEP (Holmium Laser Enucleation of the Prostate) procedure
  Interventions: Other: SOLTIVE Thulium Laser
- Control Arm: Use of Holmium Laser for HoLEP (Holmium Laser Enucleation of the Prostate) procedure
  Interventions: Other: Standard of Care (Holmium Laser)

INTERVENTIONS:
Other: SOLTIVE Thulium Laser — Use of SOLTIVE Thulium laser for HoLEP
  Groups: Solep Arm
Other: Standard of Care (Holmium Laser) — Use of Holmium laser for HoLEP
  Groups: Control Arm

SUMMARY:
To compare intraoperative as well as postoperative outcomes of SOLTIVE Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP) vs Holmium Laser Enucleation of the Prostate.

Our hypothesis is that utilizing the SOLTIVE Thulium laser enucleation of the prostate will result in a more efficient procedure, comparable results to that of Holmium laser enucleation of the prostate and subjective improvement of prior device limitations

DETAILED DESCRIPTION:
Thulium laser is continuous wave laser which offers numerous potential benefits compared to alternative lasers and surgical procedures used for BPH. The SOLTIVE Laser system is a compact system which is significantly smaller than Holmium laser systems. The laser fiber is also smaller in diameter allowing for improved maneuverability with decreased fiber degradation and endoscope damage. The continuous wave pattern produces fast, hemostatic cuts during the removal and furthermore the associated hemostasis improves the visual field. Additionally, based on the 1940nm wavelength is absorbed nearly five times more in water. For all the stated reasons, the SOLTIVE Thulium Laser should improve the enucleation efficiency and warrants further investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age or older
2. Patients must be diagnosed with benign prostatic hyperplasia
3. Patients must opt for surgical management of their BPH with laser enucleation

Exclusion Criteria:

1. Patients with a concomitant neurogenic bladder diagnosis (SCI, Parkinson, MS, cerebral palsy)
2. Patients with prostate glands greater or equal to 200 grams
3. Patients who are enrolled in other surgical or interventional trials at the time of this study are not eligible.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Study is looking at benign prostatic hypeplasia (BPH) - therefore men are the only gender to enroll. Women do not have prostates
Study Population: Patients will present to clinic for treatment of BPH assessment and evaluation per routine clinical care. Patients will be identified by clinical care team as an eligible candidate for study participation.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2022-11-30 (Actual); Study Completion 2024-05-02 (Actual)

PRIMARY OUTCOMES:
Comparing the SOLTIVE Thulium Fiber to the Holmium Laser for HoLEP | up to 1 year
  To evaluate SOLTIVE Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP) in comparison to Holmium Laser Enucleation of the Prostate through AUA Symptom Score. AUA Symptom score will be assessed using the Scale - Mild (under 7 cumulative score, moderate 8-19 score, and severe is a cumulative score over 20).

SECONDARY OUTCOMES:
Compare intraoperative components between the two surgical approaches | up to 1 year
  To compare intraoperative components of SOLTIVE Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP) vs Holmium Laser Enucleation of the Prostate
Compare post-operative outcomes of the two surgical approaches | up to 2 years
  To compare post-operative components of SOLTIVE Thulium Fiber Laser Enucleation of the Prostate (ThuFLEP)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Neff, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medcial Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No